CLINICAL TRIAL: NCT06491290
Title: Modelling of Correlation Between Emergency Department Admissions and Location-specific Air Quality and Weather in the Florence Urban Area
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Vice Director Emergency Department, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 24192_oss
Record Dates: First submitted 2024-06-21; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Emergency Service, Hospital; Air Pollution; Weather
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort
  Interventions: Other: No intervention administered

INTERVENTIONS:
Other: No intervention administered — NA (not applicable)

SUMMARY:
The goal of this observational study is to evaluate the impact of primary air pollutants and weather parameters on emergency department (ED) visits in the metropolitan area of Florence.

DETAILED DESCRIPTION:
This is a retrospective, single-center, observational cohort study aimed at investigate the impact of primary air pollutant concentrations and weather parameters on emergency department (ED) visits in the metropolitan area of Florence.

Anonymous data for each individual ED visit is retrieved from the hospital medical record. The daily concentrations of PM2.5, PM10, NO2, SO2 and O3 and the levels of atmospheric pressure, humidity and temperature are recorded by stations of the dedicated local agencies. The relationship between ED daily visits and pollutant concentrations or weather parameters are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive emergency department visits within the study period

Exclusion Criteria:

* Patients resident outside the metropolitan area investigated
* Patients admitted to the emergency department for traumatic injuries

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of consecutive patients presenting to the Emergency Departments (ED) of the participating hospital.
Sampling Method: Non-Probability Sample
Enrollment: 480000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
number of daily emergency department visits | through study completion, 1 year
  Total number of emergency department visits on a given day

OTHER OUTCOMES:
number of patients with Levels of Urgency (I-V) of emergency department visits | through study completion, 1 year
  Levels of urgency of emergency department visits defined according to the Canadian triage system. With I emergency and V non-urgent visit
Number of patients with the most frequent primary complaints of emergency department visits | through study completion, 1 year
Number of patients hospitalised | through study completion, 1 year
  Admission to a hospital ward
In-hospital mortality | through study completion, 1 year
  Death occurring either in the emergency department or following admission to ward

CONTACTS AND LOCATIONS:
Locations (1):
- SOD Medicina e Chirurgia d'Urgenza ed Accettazione, Azienda Ospedaliera-Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gnerucci A, Rossetto A, Faraoni P, Ranaldi F, Cavallaro G, Tonietti B, Santosuosso U, Bonaccorsi L, Nazerian P; SIMEU Study Group. Particulate matter concentration is associated with increased utilization of the emergency department: a single-centre time-series analysis. Intern Emerg Med. 2025 Jun 19. doi: 10.1007/s11739-025-04013-2. Online ahead of print. PMID 40537710